CLINICAL TRIAL: NCT05260619
Title: Phase II Trial of Lenalidomide Maintenance After High-dose Methotrexate-based Immunochemotherapy in Patients With Primary Central Nervous System Lymphoma
Brief Title: Lenalidomide Maintenance Treatment in Patients With Primary Central Nervous System Lymphoma
Acronym: PCNSL-LEM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Samyang BioPharm (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-2107-699-001
Record Dates: First submitted 2022-02-18; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Central Nervous System Lymphoma
MeSH Terms: interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): lenalidomide will be given as maintenance treatment to 28 PCNSL patients after achieving response to high-dose methotrexate-based immunochemotherapy
  Interventions: Drug: lenalidomide

INTERVENTIONS:
Drug: lenalidomide — Patients with MRI documented response CR or PR after induction chemotherapy will enter the study protocol of lenalidomide maintenance (at a dose of 15 mg per day, on days 1 to 21 of each 28-day cycle) for up to 12 cycles or until the patients withdrew consent, the disease progressed, or unacceptable toxic effects occurred.
  Other Names: Lenalid®

SUMMARY:
The study will include 28 patients with primary CNS DLBCL who are ineligible with autologous hematopoietic stem cell transplantation or whole brain radiation therapy as consolidation therapy.

Induction treatment will include Rituximab and high dose methotrexate protocol (containing at least methotrexate and one more chemotherapy agent).

Patients with MRI documented response CR or PR after induction chemotherapy will enter the study protocol of lenalidomide maintenance (at a dose of 15 mg per day, on days 1 to 21 of each 28-day cycle) for a maximum of 12 cycles, withdrew consent, the disease progressed, or unacceptable toxic effects occurred.

DETAILED DESCRIPTION:
The study will include 28 patients with primary CNS DLBCL who are ineligible with autologous hematopoietic stem cell transplantation or whole brain radiation therapy as consolidation therapy.

Induction treatment will include Rituximab and high dose methotrexate protocol (containing at least methotrexate and one more chemotherapy agent).

Patients with MRI documented response CR or PR after induction chemotherapy will enter the study protocol of lenalidomide maintenance (at a dose of 15 mg per day, on days 1 to 21 of each 28-day cycle) for up to 12 cycles or until the patients withdrew consent, the disease progressed, or unacceptable toxic effects occurred.

Maintenance therapy has to be started 6 weeks after the last dose of induction chemotherapy. Response evaluation by brain MRI has to be checked every 3 months after starting maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

1. PCNSL patients whose achieved response (CR/PR) after first line immunochemotherapy treatment
2. histology confirmed to be PCNSL
3. ECOG < 3
4. Hematology values must be within the following limits:

   Absolute neutrophil count (ANC) ≥ 1000/µl Platelets ≥75,000/µl
5. Biochemical values within the following limits:

   Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x upper limit of normal (ULN) Total bilirubin ≤ 2.0 x ULN Creatinine clearance (CrCl) of greater than or equal to 30 mL/min.
6. Females of childbearing potential* must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days and again within24 hours prior to prescribing lenalidomide for Cycle 1 and must either commit to continued abstinence from heterosexual intercourse or begin two acceptable methods of birth control, one highly effective method and one additional effective method at the same time, at least 28 days before she starts taking lenalidomide.

   *A female of childbearing potential is a sexually mature female who: 1) has not undergone a hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or 2) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time during the preceding 24 consecutive months).
7. Men must agree to use a latex condom during sexual contact with a female of childbearing potential even if they have had a successful vasectomy.
8. Patient must understand and voluntarily sign an informed consent form, with the understanding that the patient may withdraw consent at any time without prejudice to future medical care.

Exclusion Criteria:

1. Pregnant or breastfeeding females.
2. Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk.
3. Known history of human immunodeficiency virus (HIV) or active Hepatitis C Virus or active Hepatitis B Virus infection or any uncontrolled active systemic infection requiring intravenous (IV) antibiotics.
4. Patients with extra-central nervous system lymphoma
5. Patients who were previously exposed and who developed adverse events, hypersensitivity or desquamating rash to lenalidomide
6. prior cancer history

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 2-year
  progression-free survival

SECONDARY OUTCOMES:
ORR | 2-year
  Overall response rate
OS | 2-year
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Please Select, South Korea

IPD SHARING:
Plan to Share IPD: No